CLINICAL TRIAL: NCT05691283
Title: Right Lateralized Posterior Cerebellar tDCS in Children With Autism Spectrum Disorder
Brief Title: Cerebellar Transcranial Direct Current Stimulation (tDCS) in Children With Autism Spectrum Disorder: Raynor Cerebellum Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Tsai, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2022-0689
Record Dates: First submitted 2022-12-21; First posted 2023-01-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Children; Young adults; Autism Spectrum Disorder; Transcranial direct current stimulation; tDCS
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- transcranial direct current stimulation (tDCS), then sham stimulation (Experimental): Participants receives three weeks of 20-minute tDCS stimulation. After a washout period of 3 months, they then receive three weeks of sham stimulation
  Interventions: Device: trans cranial direct current stimulation (tDCS); Device: Sham
- Sham stimulation, then transcranial direct current stimulation (tDCS) (Experimental): Participants receives three weeks of sham stimulation. After a washout period of 3 months, they then receive three weeks of 20-minute tDCS stimulation
  Interventions: Device: trans cranial direct current stimulation (tDCS); Device: Sham

INTERVENTIONS:
Device: trans cranial direct current stimulation (tDCS) — Three weeks of 20-minute tDCS stimulation
Device: Sham — Three weeks of sham stimulation

SUMMARY:
The purpose of this research study is to investigate the effects of transcranial direct current stimulation (tDCS) on some of the challenges faced by children with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
The study will be randomized, double-blind, within subject crossover design. It will involve a group of 30-40 children and young adults with Autism Spectrum Disorder (ASD). We may recruit up to 60 subjects. Diagnosis of ASD will be confirmed with the Autism Diagnostic Interview-Revised (ADI-R) or Autism Diagnostic Observation Schedule-2 (ADOS-2) by a research-reliable clinician. Each participant will undergo a sham condition and a transcranial direct current stimulation (tDCS) condition, the order of sham and tDCS conditions will be randomly assigned to each participant during baseline testing. Sham refers to participants only receiving 1 milliamp of tDCS stimulation for 1 minute, and tDCS stimulation refers to 20 minutes of tDCS stimulation. The study involves an initial screening visit followed by two sessions with three months between each session period. Each session includes the following: pre-testing and imaging, tDCS 3-week session, post-testing and imaging. Participants will complete an initial screening to confirm clinical diagnosis of ASD, determine baseline cognitive functioning, and complete a practice Magnetic Resonance Imaging (MRI) and Magnetoencephalography (MEG) session. At pre-testing, they will complete a psychometric battery, as well as undergo safety screening, and an MRI and/or MEG. Each 3-week tDCS sessions will be randomized, and each participant will undergo three weeks of sham stimulation and three weeks of 20-minute tDCS stimulation. Neither the researchers nor the participants will know which group they are assigned during each three-week session.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5 to 21, male and female, with known autism spectrum disorder as diagnosed by a clinician

Exclusion Criteria:

* Pregnancy
* Brain implants
* Pacemakers
* Any biomedical or metal implants in any part of body
* Hearing or visual impairment
* History of brain injury
* Known brain or skull abnormality other than those that may be associated with ASD

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Social behavior as measured by Reading the Mind in the Eyes (RME) Child Version | Baseline
  Reading the Mind in the Eyes (RME) Child Version will be used to measure complex mental state recognition. This test consists of 28 photographs of the eye region of the human face, each surrounded by four words. Participants pick the word that best describes what the person in the photo is thinking or feeling. Scores range from 0-28, higher score indicates very accurate at decoding a person's facial expressions around their eyes.
Social behavior as measured by Reading the Mind in the Eyes (RME) Child Version | Post Treatment (approx at 3 month)
  Reading the Mind in the Eyes (RME) Child Version will be used to measure complex mental state recognition. This test consists of 28 photographs of the eye region of the human face, each surrounded by four words. Participants pick the word that best describes what the person in the photo is thinking or feeling. Scores range from 0-28, higher score indicates very accurate at decoding a person's facial expressions around their eyes.
Social behavior as measured by Cyberball/Social Ball Throwing Task | Baseline
  Cyberball/Social Ball Throwing Task will be used to measure social interaction. In this task, the participant engaged in a virtual ball throwing game with two other players. There are three conditions the participants will be randomly assigned to. In two conditions participants are thrown the ball an equal number of times, in the other condition the participant is only thrown the ball a few times. After the participant completes the task, they are given a rating scale to rate how well they trust and prefer the other two players on a scale from 1-7 (totally mistrust to totally trust). The ratings indicated how well the subject was able to determine if they were left out of the group"
Social behavior as measured by Cyberball/Social Ball Throwing Task | Post Treatment (approx at 3 month)
  Cyberball/Social Ball Throwing Task will be used to measure social interaction. In this task, the participant engaged in a virtual ball throwing game with two other players. There are three conditions the participants will be randomly assigned to. In two conditions participants are thrown the ball an equal number of times, in the other condition the participant is only thrown the ball a few times. After the participant completes the task, they are given a rating scale to rate how well they trust and prefer the other two players on a scale from 1-7 (totally mistrust to totally trust). The ratings indicated how well the subject was able to determine if they were left out of the group"
Sensorimotor behavior as measured by Grip Strength | Baseline
  Participants grip a specially designed fiber optic device (Aither Engineering, Inc.). This device detects nanometer changes in grip force which are calibrated in Newtons. Participants are instructed to rest their arm in a relaxed position. Subjects use their thumb and index finger to press against grip device. Prior to testing, each subject will complete the maximum voluntary contraction for each hand during trials of 3 seconds each with 15 seconds in between each trial. The subject is then instructed to press as hard as they can when the screen says "go" using only the thumb and pointer finger.
Sensorimotor behavior as measured by Grip Strength | Post Treatment (approx at 3 month)
  Participants grip a specially designed fiber optic device (Aither Engineering, Inc.). This device detects nanometer changes in grip force which are calibrated in Newtons. Participants are instructed to rest their arm in a relaxed position. Subjects use their thumb and index finger to press against grip device. Prior to testing, each subject will complete the maximum voluntary contraction for each hand during trials of 3 seconds each with 15 seconds in between each trial. The subject is then instructed to press as hard as they can when the screen says "go" using only the thumb and pointer finger.
Sensorimotor behavior as measured by Reach Task | Baseline
  Participants will be positioned at a table with reaching arm resting on the table in a neutral position. The task includes picking up small objects placed on the table and placing the objects one by one into a target container in two trials: preferred and non-preferred hands. The task is rated on a 6-point rating scale, where 5 represents weakest performance, and 0 represents best performance. Each item is given a raw score and a standard score, which translate to a component score and percentile rank.
Sensorimotor behavior as measured by Reach Task | Post Treatment (approx at 3 month)
  Participants will be positioned at a table with reaching arm resting on the table in a neutral position. The task includes picking up small objects placed on the table and placing the objects one by one into a target container in two trials: preferred and non-preferred hands. The task is rated on a 6-point rating scale, where 5 represents weakest performance, and 0 represents best performance. Each item is given a raw score and a standard score, which translate to a component score and percentile rank.
Sensorimotor behavior as measured by Sensory Profile-2 | Baseline
  A parent self-report form designed to assess sensory processing patterns in children and adolescents. The report includes three subscales: sensory system, behavior, and sensory pattern.Each item is scored on a Likert scale from 1 to 5 (1=Much Less Than Others, 2=Less Than Others, 3=Just Like the Majority of Others, 4=More Than Others, 5=Much More Than Others). Raw scores are totaled and converted to percentile ranks based on participant age.
Sensorimotor behavior as measured by Sensory Profile-2 | Post Treatment (approx at 3 month)
  A parent self-report form designed to assess sensory processing patterns in children and adolescents. The report includes three subscales: sensory system, behavior, and sensory pattern.Each item is scored on a Likert scale from 1 to 5 (1=Much Less Than Others, 2=Less Than Others, 3=Just Like the Majority of Others, 4=More Than Others, 5=Much More Than Others). Raw scores are totaled and converted to percentile ranks based on participant age.
Neurophysiological impacts as measured by Magnetoencephalography (MEG) | Baseline
  MEG data will be processed using AFNI (https://afni.nimh.nih.gov/). Using all channels of the MEG data, strength and latency of responses are measured by transforming each subject's raw MEG activity into brain space. A spatial filter is applied which separates the source activity from different brain regions to observe overlap at the sensor level. This analysis will assess functional connectivity between the region of interest (ROI) voxel, the right Crus I of the cerebellum, compared to all other voxels in the brain. Seed-based voxel correlation analysis enables researchers to see the statistical correlation between the ROI activity and activity in other cortical areas. This correlation reveals patterns of connectivity between the ROI and other cortical regions. The second level analysis will utilize a one-way ANOVAs will compare baseline measures (Cyberball, Precision Grip) and demographics (e.g. age) within groups. The within subjects' effect of tDCS on task scores will be evaluated
Neurophysiological impacts as measured by Magnetoencephalography (MEG) | Post Treatment (approx at 3 month)
  MEG data will be processed using AFNI (https://afni.nimh.nih.gov/). Using all channels of the MEG data, strength and latency of responses are measured by transforming each subject's raw MEG activity into brain space. A spatial filter is applied which separates the source activity from different brain regions to observe overlap at the sensor level. This analysis will assess functional connectivity between the region of interest (ROI) voxel, the right Crus I of the cerebellum, compared to all other voxels in the brain. Seed-based voxel correlation analysis enables researchers to see the statistical correlation between the ROI activity and activity in other cortical areas. This correlation reveals patterns of connectivity between the ROI and other cortical regions. The second level analysis will utilize a one-way ANOVAs will compare baseline measures (Cyberball, Precision Grip) and demographics (e.g. age) within groups. The within subjects' effect of tDCS on task scores will be evaluated
Neurophysiological impacts as measured by functional magnetic resonance imaging (fMRI) | Baseline
  fMRI data will be processed using AFNI (https://afni.nimh.nih.gov/). A regression analyses is used (3dDeconvolve and 3dREML) for each subject. Data collected from MRI acquisition will be analyzed at two levels. The first level of analysis will use seed-based voxel correlational analysis, a statistical technique for observing differences in brain activity. This analysis will assess functional connectivity between the region of interest (ROI) voxel, the right Crus I of the cerebellum, compared to all other voxels in the brain. Seed-based voxel correlation analysis enables researchers to see the statistical correlation between the ROI activity and activity in other cortical areas. This correlation reveals patterns of connectivity between the ROI and other cortical regions. The second level analysis will utilize a one-way ANOVAs will compare baseline measures (Cyberball, Precision Grip) and demographics (e.g. age) within groups.
Neurophysiological impacts as measured by functional magnetic resonance imaging (fMRI) | Post Treatment (approx at 3 month)
  fMRI data will be processed using AFNI (https://afni.nimh.nih.gov/). A regression analyses is used (3dDeconvolve and 3dREML) for each subject. Data collected from MRI acquisition will be analyzed at two levels. The first level of analysis will use seed-based voxel correlational analysis, a statistical technique for observing differences in brain activity. This analysis will assess functional connectivity between the region of interest (ROI) voxel, the right Crus I of the cerebellum, compared to all other voxels in the brain. Seed-based voxel correlation analysis enables researchers to see the statistical correlation between the ROI activity and activity in other cortical areas. This correlation reveals patterns of connectivity between the ROI and other cortical regions. The second level analysis will utilize a one-way ANOVAs will compare baseline measures (Cyberball, Precision Grip) and demographics (e.g. age) within groups.

SECONDARY OUTCOMES:
Executive functioning as measured by Flanker Inhibitory Control and Attention | Baseline
  The NIH Toolbox Flanker Inhibitory Control and Attention Test measures both a participant's attention and inhibitory control. Accuracy and reaction scores range in value between 0 and 5. If accuracy scores for the participant reach more than 80%, the reaction time score and accuracy score are combined. Combined scores range in value from 0-10. This score shows how accurate and how quickly the subject responded, the high the score the more accurate and quickly each subject responded.
Executive functioning as measured by Flanker Inhibitory Control and Attention | Post Treatment (approx at 3 month)
  The NIH Toolbox Flanker Inhibitory Control and Attention Test measures both a participant's attention and inhibitory control. Accuracy and reaction scores range in value between 0 and 5. If accuracy scores for the participant reach more than 80%, the reaction time score and accuracy score are combined. Combined scores range in value from 0-10. This score shows how accurate and how quickly the subject responded, the high the score the more accurate and quickly each subject responded.
Executive functioning as measured by Dimensional Card Change Sort | Baseline
  The Dimensional Change Card Sort (DCCS) is a measure of cognitive flexibility, also known as task switching or set shifting. Scoring is based on a combination of accuracy and reaction time. Accuracy and reaction scores range in value between 0 and 5. If accuracy scores for the participant reach more than 80%, the reaction time score and accuracy score are combined. Combined scores range in value from 0-10. This score shows how accurate and how quickly the subject responded, the high the score the more accurate and quickly each subject responded.
Executive functioning as measured by Dimensional Card Change Sort | Post Treatment (approx at 3 month)
  The Dimensional Change Card Sort (DCCS) is a measure of cognitive flexibility, also known as task switching or set shifting. Scoring is based on a combination of accuracy and reaction time. Accuracy and reaction scores range in value between 0 and 5. If accuracy scores for the participant reach more than 80%, the reaction time score and accuracy score are combined. Combined scores range in value from 0-10. This score shows how accurate and how quickly the subject responded, the high the score the more accurate and quickly each subject responded.
Working memory as measured by Stanford Binet-V Working Memory Subtest | Baseline
  Stanford Binet-V Working Memory Subtest assesses how well the subject recalls facts and objects. This area assesses how well the subject recalls facts and objects. At lower levels, the non-verbal test involves asking the subject to find an object hidden under a cup, or block tapping in which the subject must repeat a sequence of tapping on blocks initiated by the examiner. The verbal test requires the subject to recall the last words of several sentences in a series. Raw scores are the total number of items correct and are converted into standard scores (0-119) for each subtest based on participant age. Standard scores of 100-110 are considered average for the subjects age range
Working memory as measured by Stanford Binet-V Working Memory Subtest | Post Treatment (approx at 3 month)
  Stanford Binet-V Working Memory Subtest assesses how well the subject recalls facts and objects. This area assesses how well the subject recalls facts and objects. At lower levels, the non-verbal test involves asking the subject to find an object hidden under a cup, or block tapping in which the subject must repeat a sequence of tapping on blocks initiated by the examiner. The verbal test requires the subject to recall the last words of several sentences in a series. Raw scores are the total number of items correct and are converted into standard scores (0-119) for each subtest based on participant age. Standard scores of 100-110 are considered average for the subjects age range

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tsai, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dalls, Texas, United States

IPD SHARING:
Plan to Share IPD: No